CLINICAL TRIAL: NCT03691818
Title: A Phase 2, Multicenter, Double-blind and Placebo and Active Control Study to Evaluate the Initial Efficacy and Safety of X0002 Spray in Treatment of Subjects With Osteoarthritis of the Knee
Brief Title: Evaluate Efficacy and Safety of X0002 in Treatment of Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin XinChen-Techfields Pharma Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TFR-X0002-201
Record Dates: First submitted 2018-09-03; First posted 2018-10-02 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-01

CONDITIONS: KNEE OSTEOARTHRITIS
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Drug Evaluation; Ibuprofen; Bulk Drugs

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Low-dose test drug group (Experimental): X0002 Spray 1 Spray/time/Knee, 2 times/day; Ibuprofen Placebo Tab 400 mg/time, 3 times /day.
  Interventions: Drug: X0002 Spray; Drug: Ibuprofen Placebo Tab
- Low-dose active drug control group (Active Comparator): Ibuprofen Tablet 400 mg/time, 3 times /day; X0002 Placebo Spray 1 Spray/time/Knee, 2 times/day.
  Interventions: Drug: Ibuprofen Tablet; Drug: X0002 Placebo Spray
- Low-dose placebo control group (Placebo Comparator): Placebo Spray 1 Spray/time/Knee, 2 times/day; Ibuprofen Placebo Tab 400 mg/time, 3 times/day.
  Interventions: Drug: Ibuprofen Placebo Tab; Drug: X0002 Placebo Spray
- Medium-dose test drug group (Experimental): X0002 Spray 2 Spray/time/Knee, 2 times/day; Ibuprofen Placebo Tab 400 mg/time, 3 times /day.
  Interventions: Drug: X0002 Spray; Drug: Ibuprofen Placebo Tab
- Medium-dose active drug control group (Active Comparator): X0002 Placebo Spray 2 Spray/time/Knee, 2 times/day; Ibuprofen Tablet 400 mg/time, 3 times /day.
  Interventions: Drug: Ibuprofen Tablet; Drug: X0002 Placebo Spray
- Medium-dose placebo control group (Placebo Comparator): X0002 Placebo Spray 2 Spray/time/Knee, 2 times/day; Ibuprofen Placebo Tab 400 mg/time, 3 times /day.
  Interventions: Drug: Ibuprofen Placebo Tab; Drug: X0002 Placebo Spray
- High-dose test drug group (Experimental): X0002 Spray 4 Spray/time/Knee, 2 times/day; Ibuprofen Placebo Tab 400 mg/time, 3 times /day.
  Interventions: Drug: X0002 Spray; Drug: Ibuprofen Placebo Tab
- High-dose active drug control group (Active Comparator): X0002 Placebo Spray 4 Spray/time/Knee, 2 times/day; Ibuprofen Tablet 400 mg/time, 3 times /day.
  Interventions: Drug: Ibuprofen Tablet; Drug: X0002 Placebo Spray
- High-dose placebo control group (Placebo Comparator): X0002 Placebo Spray 4 Spray/time/Knee, 2 times/day; Placebo Tablet 400 mg/time, 3 times /day.
  Interventions: Drug: Ibuprofen Placebo Tab; Drug: X0002 Placebo Spray

INTERVENTIONS:
Drug: X0002 Spray — According to the different dose groups assigned, each knee joint was sprayed with 1, 2 or 4 sprays.
  Other Names: Test drug
  Arms: High-dose test drug group; Low-dose test drug group; Medium-dose test drug group
Drug: Ibuprofen Tablet — Ibuprofen Tab 400mg, tid.
  Other Names: Active drug
  Arms: High-dose active drug control group; Low-dose active drug control group; Medium-dose active drug control group
Drug: Ibuprofen Placebo Tab — Ibuprofen Placebo Tab 400mg, tid.
  Other Names: Placebo Oral Tablet
  Arms: High-dose placebo control group; High-dose test drug group; Low-dose placebo control group; Low-dose test drug group; Medium-dose placebo control group; Medium-dose test drug group
Drug: X0002 Placebo Spray — According to the different dose groups assigned, each knee joint was sprayed with 1, 2 or 4 sprays.
  Other Names: Placebo Spray
  Arms: High-dose active drug control group; High-dose placebo control group; Low-dose active drug control group; Low-dose placebo control group; Medium-dose active drug control group; Medium-dose placebo control group

SUMMARY:
This study is a randomized, double-blind clinical trial in a Chinese population.

DETAILED DESCRIPTION:
This study is a randomized, double-blind clinical trial in a Chinese population. Active drug and placebo were used as controls to observe the relative efficacy of X0002 spray.

ELIGIBILITY:
Inclusion Criteria:

* 1. Ability to read and provide written, personally signed, and dated informed consent to participate in the study, in accordance with the GCP and applicable regulations, before completing any study related procedures.

  2. An understanding, ability, and willingness to fully comply with study procedures and restrictions.

  3. Subject must be a male or female between 40 and 75 years of age, inclusive.

  4. Female subjects must either not be of childbearing potential (defined as postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy, or hysterectomy]) or be willing to practice at least 1 of the following medically acceptable methods of birth control: Hormonal methods such as oral, implantable, injectable, vaginal ring, or transdermal contraceptives for a minimum of 1 full cycle (based on the subjects usual menstrual cycle period) before study drug administration.
  1. Intrauterine device.
  2. Double-barrier method (condoms, sponge, or diaphragm with spermicidal jellies or cream).

     5. Subject must have a diagnosis of idiopathic OA according to the American College of Rheumatology clinical and radiographic criteria, and fulfillment of at least four of the 6 criteria: age of ≥50 years stiffness lasting <30 minutes after getting up in the morning crepitus Bone tenderness Bone enlargement No joint fever

     6. Subject must have a history of clinically symptomatic OA of the knee for ≥6 months.

     7. Subject must have had knee pain while standing, walking, and/or in motion for at least 14 days during the month prior to screening.

     8. Subject must have a knee pain score ≥40 mm and <90 mm on a 100 mm VAS (without analgesic medication) on at least 7 of the 10 days prior to randomization(according to the subject's diary card records).

     9. Subject must have a WOMAC pain average score of knee ≥40 mm and <90 mm starting on the first screening visit.

     10. Subject must be willing to discontinue any NSAIDs or other analgesic (e.g. aspirin) or potentially confounding concomitant treatments (e.g. physiotherapy, acupuncture) starting on the first screening visit until completing participation in the study. (The use of ≤325 mg acetylsalicylic acid per day as cardiac prophylaxis is permitted.) The subject will be allowed to take rescue medication (acetaminophen) for pain during the study except during the 24 hours prior to the Second Screening Visit, Baseline (Day1), Week 2, Week 4, Week 8, Week 12, Week 14.

     11. Subject must be willing to discontinue applying any topical preparations containing Vitamin A acids [including all trans-retinoic-acid (tretinoin), 13-cis-retinoic-acid (isotretinoin), 9-cis-retinoic-acid (alitretinoin), vitamin A (retinol), retinal, and their derivatives] to the lower limbs starting on the first screening visit until completing participation in the study. (Topical preparations containing Vitamin A acids or retinol may be applied to areas of the skin above the waist, but should not be applied to areas of the skin exposed to study medication.) 12. Subject must be willing to avoid unaccustomed physical activity (e.g. starting a new weight lifting routine) for the duration of the study starting on the first screening visit.

     13. With the exception of OA of the knee, the subject must be in good general health with no clinically significant findings from medical history, vital signs, physical examination, ECG, and routine laboratory tests that could interfere with subject safety, or pain and functional assessments, as determined by the Investigator.

     Exclusion Criteria:
* 1. The subject had a history of trauma, and the injury affected the knee joint.

  2. Subject who has secondary OA of the knee or OA of lower limb joints other than the knee that in the opinion of the Investigator, could interfere with pain and functional assessments related to the knee.

  3. Subject who has a history of total or partial knee replacement, arthroplasty, or other knee surgery on either knee.

  4. Subject who has had significant injury, as estimated by the Investigator, involving the target knee within the 6 months before screening.

  5. Subject who has skin lesions or wounds on or near the knees to be treated at Screening or on Day 1 prior to the first administration of study medication.

  6. Subject who has used opiates or corticosteroids within 30 days before screening for the target knee or who requires treatment with chronic opiates or corticosteroids.

  7. Subject who has had intra articular injections of corticosteroids, hyaluronic acid, or viscosupplements (e.g. Synvisc®) to a knee to be treated within the 3 months before screening.

  8. Subject who has a history of significant hypersensitivity, intolerance, or allergy to ibuprofen, any NSAIDs, aspirin, or acetaminophen.

  9. Subject who has had an active peptic ulceration in the 6 months prior to screening or a history of gastrointestinal (GI) bleeding within 5 years of screening.

  10. Subject who has used an anticoagulant (except aspirin up to 325 mg/day for cardiac prophylaxis) in the month prior to Screening.

  11. Subject who has positive results on fecal occult blood testing at screening or on Day 1 prior to the first administration of study medication.

  12. Subject who has a history of chronic inflammatory disease (such as rheumatoid arthritis, psoriatic arthritis, gouty arthritis), fibromyalgia, or other conditions that may affect the target joint or the functional and pain assessments (e.g. osteonecrosis, chondrocalcinosis).

  13. Subject is an asthmatic requiring treatment with systemic corticosteroids. Asthmatic subjects using inhaled corticosteroids are eligible.

  14. Subject has any clinically significant unstable cardiac, respiratory, neurological, immunological, hematological, or renal disease, or any other condition that, in the investigators opinion, could compromise the subjects welfare, ability to communicate with the study staff, or otherwise contraindicate study participation.

  15. Subject has a significant renal or hepatic disease, as indicated by clinical laboratory assessment,defined as
  1. aspartate aminotransferase, alanine aminotransferase, and lactate dehydrogenase≥3 × the upper limit of normal
  2. creatinine ≥1.5 × ULN
  3. hemoglobin<10g/dL.

     16. Subject has any other clinically significant laboratory finding at Screening that in the investigators opinion contraindicates study participation.

     17. Subject is receiving systemic chemotherapy, has an active malignancy of any type, or has been diagnosed with cancer within 5 years before Screening (excluding squamous or basal cell carcinoma of the skin).

     18. Subject has clinically significant abnormality on 12-lead ECG, including a QTc interval >450 msecs for males and 470 msecs for females.

     19. Subject has uncontrolled hypertension defined as systolic blood pressure >170 mmHg and diastolic blood pressure >90 mmHg at baseline (may be repeated after 5 minutes rest to verify).

     20. Subject is female and pregnant, planning to become pregnant during the study, or nursing.

     21. Subject participated in a previous clinical study with bromine hydrochloride spray.

     22. Subjects with known alcohol or other substance abuse.

     23. Subject participated in any other clinical trial within the past 3 months or 5 half-lives, whichever is longer.

     24. Subject is a participating Investigator, sub-investigator, study coordinator, or employee of a participating Investigator, or is an immediate family member of the aforementioned.

     25. Any factor, which in the opinion of the Investigator would jeopardize the evaluation or safety or be associated with poor adherence to the protocol.

     26. Subjects without access to telephone and/or ability to gain technology access.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Change of the Subject's Target OA Knee Compared to the Baseline as Assessed by WOMAC | week 12
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) has been used to assess subjects with OA of the hip or knee and consists of 24 questions in subscales measuring 3 concepts: pain, stiffness, and physical function. These questions measure the amount of pain, degree of difficulty in completing various day-to-day activities, and stiffness experienced in the hip or knee. Usually subject self-administered. A single question has 100 grades, where 0 = very good and 100 = very much worse. VAS (visual analog scale) scale is used for score record.
  Data for the exploratory efficacy endpoints will be summarized using descriptive statistics.
  Safety analyses will be conducted on the SAS. Safety parameters will be listed and summarized using standard descriptive statistics.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events of X0002 Spray | week 1 to week 14
  A sensitivity analysis will also be conducted on the Primary Efficacy Endpoint using an ANCOVA with treatment as a fixed class effect and WOMAC baseline pain subscale score as covariates, but the comparisons of interest will be the difference between the active and placebo subjects within each treatment group.
  The Secondary Efficacy Endpoints, change from Baseline in the WOMAC subscale scores for pain, stiffness, and functional ability, and overall WOMAC score, will be by analyzed using the same methods as the for the Primary Efficacy Endpoint.
  Safety analyses will be conducted on the SAS. Safety parameters will be listed and summarized using standard descriptive statistics, as appropriate. No formal statistical analyses are planned.
Relief of Knee Pain in Subjects With Osteoarthritis (OA) of the Knee as Evaluated by WOMAC Subscale | week 2，4，8
  The WOMAC pain subscale has 5 questions. Usually subject self-administered. A single question has 100 grades, where 0 = no pain and 100 = pain as bad as can be.
  The Primary Efficacy Endpoint is change from Baseline in the WOMAC (VAS) pain subscale score for the target knee at week 2, 4, 8, and will be analyzed by an analysis of covariance (ANCOVA). Treatment will be included as a fixed class effect and WOMAC Baseline pain subscale score as covariates.
Relief of Joint Stiffness After Using X0002 Spray as Evaluated by WOMAC Subscale | week 2，4，8, 12
  The WOMAC stiffness subscale has 2 questions. Usually subject self-administered. A single question has 100 grades, where 0 = no stiffness and 100 = stiffness as bad as can be.
  A sensitivity analysis will also be conducted on the Primary Efficacy Endpoint using an ANCOVA with treatment as a fixed class effect and WOMAC baseline stiffness subscale score as covariates, but the comparisons of interest will be the difference between the active and placebo subjects within each treatment group.
  The Secondary Efficacy Endpoints, change from Baseline in the WOMAC subscale scores for stiffness at 2, 4, 8, and 12 weeks of treatment, will be by analyzed using the same methods as the for the Primary Efficacy Endpoint.
  Safety analyses will be conducted on the SAS. Safety parameters will be listed and summarized using standard descriptive statistics, as appropriate. No formal statistical analyses are planned.
Difficulty Performing Daily Activities of OA Subjects as Assessed by WOMAC subscale | week 2，4，8, 12
  The WOMAC physical function subscale has 17 questions. Usually subject self-administered. A single question has 100 grades, where 0 = very good and 100 = very much worse.
  A sensitivity analysis will also be conducted on the Primary Efficacy Endpoint using an ANCOVA with treatment as a fixed class effect and WOMAC baseline pain subscale score as covariates, but the comparisons of interest will be the difference between the active and placebo subjects within each treatment group.
  The Secondary Efficacy Endpoints, change from Baseline in the WOMAC subscale scores for pain, stiffness, and functional ability, and overall WOMAC score at 2, 8, and 12 weeks of treatment, will be by analyzed using the same methods as the for the Primary Efficacy Endpoint.
  Safety analyses will be conducted on the SAS. Safety parameters will be listed and summarized using standard descriptive statistics, as appropriate. No formal statistical analyses are planned.
Total Score of WOMAC Subscale as Estimated by Visual Analog Scale | week 2，4，8, 12
  The WOMAC subscale has 24 questions. Usually subject self-administered. A single question has 100 grades, where 0 = very good and 100 = very much worse. The total score is 2400, the lower, the better; higher score means worse condition.
  Data for the exploratory efficacy endpoints will be summarized using descriptive statistics.
  Safety analyses will be conducted on the SAS. Safety parameters will be listed and summarized using standard descriptive statistics, as appropriate. No formal statistical analyses are planned.
Subject's Global Assessment of Disease Status of the Target Knee as Estimated by Visual Analog Scale at 2, 4, 8 and 12 Weeks of Treatment | week 2，4，8, 12
  The subject's overall evaluation of the condition is the relevant questionnaire (0-100mm visual analogue scale), which needs to be completed at the time points listed in the study flow chart. On the scale line of 100mm VAS, mark the left side to indicate "very good" and mark the right side means "Very bad." Data for the exploratory efficacy endpoints will be summarized using descriptive statistics.
  Safety analyses will be conducted on the SAS. Safety parameters will be listed and summarized using standard descriptive statistics, as appropriate. No formal statistical analyses are planned.
Subject's Global Assessment of Response to Therapy of the Target Knee as Estimated by Visual Analog Scale at 2, 4, 8 and 12 Weeks of Treatment | week 2，4，8, 12
  The subjects' overall evaluation of treatment response is that they fill in the relevant questionnaire VAS (visual analog scale) (VAS, 0~4 points), which should be completed in the time points listed in the study flow chart. 0 = very poor; 4 = very good.
  Data for the exploratory efficacy endpoints will be summarized using descriptive statistics.
  Safety analyses will be conducted on the SAS. Safety parameters will be listed and summarized using standard descriptive statistics, as appropriate. No formal statistical analyses are planned.
Amount of Rescue Medication (Acetaminophen) Consumed Per Day for Target Knee Pain | week 2，4，8, 12
  Data for the exploratory efficacy endpoints will be summarized using descriptive statistics.
  Safety analyses will be conducted on the SAS. Safety parameters will be listed and summarized using standard descriptive statistics, as appropriate. No formal statistical analyses are planned.
Pharmacokinetic parameters(Maximum Plasma Concentration [Cmax]) of X0002 | 1 h pre-dose, 1±0.5 h post-dose, 3±0.5 h post-dose, 5±0.5 h post-dose at week 8; 1 h pre-dose, 2±0.5 h post-dose, 4±0.5 h post-dose, 6±0.5 h post-dose at week 12
  Cmax of X0002 will be calculated.
Pharmacokinetic parameters(Area Under Curve [AUC]) of X0002 | 1 h pre-dose, 1±0.5 h post-dose, 3±0.5 h post-dose, 5±0.5 h post-dose at week 8; 1 h pre-dose, 2±0.5 h post-dose, 4±0.5 h post-dose, 6±0.5 h post-dose at week 12
  AUC of X0002 will be calculated.

OTHER OUTCOMES:
Investigator's Global Assessment of Subjects' Disease Status and Therapy Effects at 2, 4, 8 and 12 Weeks of Treatment | week 2，4，8, 12
  The researchers used the visual analog scale (VAS) for the overall assessment of the disease (VAS scales, 0~4 points), which needed to be completed at the time points listed in the study flow chart. 0 = very poor; 4 = very good.
  Data for the exploratory efficacy endpoints will be summarized using descriptive statistics.
  Safety analyses will be conducted on the SAS. Safety parameters will be listed and summarized using standard descriptive statistics, as appropriate. No formal statistical analyses are planned.
Change in the WOMAC Subscale Scores for Pain, Stiffness and Functional Ability of Target Knee | week 14
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) has been used to assess subjects with OA of the hip or knee and consists of 24 questions in subscales measuring 3 concepts: pain, stiffness, and physical function. These questions measure the amount of pain, degree of difficulty in completing various day-to-day activities, and stiffness experienced in the hip or knee. Usually subject self-administered. A single question has 100 grades, where 0 = very good and 100 = very much worse.
  Change in the WOMAC subscale scores for pain, stiffness, and functional ability at week 14 of treatment, will be by analyzed using the same methods as the for the Primary Efficacy Endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Zeng Xiaofeng, Principal Investigator — lead institution
Locations (1):
- Chinese Academy of Medical Science & Peking Union Medical college Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No